CLINICAL TRIAL: NCT05979038
Title: Evaluation of the Effect of Metformin on the Clinical Outcome of ICU Patients With Sepsis
Brief Title: Clinical Evaluation of the Effect of Metformin in Sepsis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: German University in Cairo (Other)
Responsible Party: Principal Investigator, Mai Tarek Ghannoum, Assistant Lecturer of Clinical Pharmacy, German University in Cairo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FMASU MD146/2023
Record Dates: First submitted 2023-07-30; First posted 2023-08-07 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis | interventions — Metformin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Metformin arm (Experimental): In this arm patients will administrate metformin 500 mg three times a day together with the standard care of sepsis.
  Interventions: Drug: Metformin
- Control Arm (No Intervention): In this arm patients will receive the standard care of sepsis only

INTERVENTIONS:
Drug: Metformin — Patients in the intervention arm will take metformin 500mg three times a day
  Other Names: Glucophage
  Arms: Metformin arm

SUMMARY:
Sepsis is defined as life-threatening organ dysfunction caused by a dysregulated host response to infection. It is considered a condition that arises when the body's response to an infection injures its own tissues and organs. The pathogenesis of sepsis is very complicated as it involves imbalance in inflammatory response, immune dysfunction, mitochondrial damage, coagulopathy, neuroendocrine immune network abnormalities, endoplasmic reticulum stress, autophagy, and other pathophysiological processes, and leads to organ dysfunction. Inflammatory Imbalance represents the most critical basis of sepsis pathogenesis. Sepsis is associated with many biochemical abnormalities that is correlated with patients' prognosis and risk of mortality including increased levels of lactate, procalcitonin and inflammatory cytokines as TNF alpha.

Metformin is an oral anti-diabetic drug from the class of biguanides. It is the first line treatment of diabetes type 2. It is widely used as it has good safety profile, low side effect and cheap cost. Metformin has been reported to have an anti-inflammatory and anti-microbial effect.

Some studies have shown that metformin has a beneficial effect in sepsis patients. Our study will be the first prospective controlled randomized trial to assess the clinical outcome of metformin in patients with sepsis.

DETAILED DESCRIPTION:
Sepsis is defined as life-threatening organ dysfunction caused by a dysregulated host response to infection. It is considered a life-threatening condition that arises when the body's response to an infection injures its own tissues and organs (Singer et al., 2016a). Organ dysfunction can be defined as an increase in the Sequential (sepsis related) Organ Failure Assessment (SOFA) score more than two points consequent to the infection. A SOFA score more than two points indicates that an overall mortality risk of approximately 10% in hospital population with suspected infection.(Singer et al., 2016b). Septic shock is defined as subset of sepsis in which circulatory, cellular, and metabolic abnormalities are associated with a greater risk of mortality than sepsis alone. Patients with septic shock can be identified with a clinical construct of sepsis with persisting hypotension requiring vasopressors to maintain MAP (mean arterial pressure) more than or equal 65mmHg and having a serum lactate level >2 mmol/L (18mg/dL) despite adequate volume resuscitation (Seymour et al., 2016).

Sepsis and septic shock are major healthcare problems, affecting millions of people around the world each year with a mortality rate between one in three and one in six of those it affects (Evans et al., 2021). According to a meta-analysis conducted in 2020, it was found that the incidence of sepsis was 189 hospital-treated sepsis cases per 100,000 person-years with a 26.7% mortality rate. In ICU patients, the incidence was 58 per 100,000 person-years with a mortality rate of 41.9% prior to hospital discharge (Fleischmann-Struzek et al., 2020).

The pathogenesis of sepsis is very complicated as it involves imbalance in inflammatory response, immune dysfunction, mitochondrial damage, coagulopathy, neuroendocrine immune network abnormalities, endoplasmic reticulum stress, autophagy, and other pathophysiological processes, and leads to organ dysfunction. Inflammatory Imbalance represents the most critical basis of sepsis pathogenesis. The host's initial acute response to invasive pathogens causes macrophages to engulf the pathogens and produce a range of pro-inflammatory cytokines, and this can trigger cytokine storms and activate the innate immune system. The activation of the innate immune system is mediated by pattern-recognition receptors (PRRs), which initiate a series of activation in immune cells by detecting damage-associated molecular patterns (DAMPs) or pathogen-associated molecular patterns (PAMPs), and thus upregulate the expression of inflammation related genes. In the immune response to sepsis, both exogenous factors derived from the pathogen (e.g., lipopolysaccharide (LPS)) and endogenous factors released by injured cells (e.g., high-mobility group box-1 (HMGB-1) protein) can interact with various PRRs, such as Toll-like receptors (TLRs), which leads to the activation of several pathways including p38 mitogen-activated protein kinase (MAPK), and nuclear factor-κB (NF-κB) signaling pathways. These events are followed by the production of inflammatory cytokines such as interleukin (IL)-1, IL-6, tumor necrosis factor-α (TNF-α), interferon (IFN) regulatory factor 7 (IRF7), and adaptor protein 1 (AP-1) (Huang, Cai and Su, 2019).

Moreover, studies have also shown that in early stages of sepsis, exaggerated endothelial activation, vascular leakage, disturbance of blood flow, as well as other derangements cause the loss of vascular integrity, which contributes significantly to sepsis-associated organ failure. Therapies interfering endothelial activation are potential to attenuate sepsis-induced organ dysfunction (Tian et al., 2019) Sepsis is associated with many biochemical abnormalities that is correlated with patients' prognosis and risk of mortality including increased levels of lactate, procalcitonin and inflammatory cytokines as TNF alpha.(Cho and Choi, 2014) Despite great efforts was done to understand the pathogenesis of sepsis and investigate therapeutic strategies, the management of sepsis remains a clinical challenge (Tian et al., 2019). Till current date the pathogenesis of sepsis is not completely clear but most of the studies suggested that the release of inflammatory factors by patient's innate immune cell plays an important role in the disease progression (Liang et al., 2019). Recently several studies revealed the anti-inflammatory effect of some drugs in sepsis. One of the drugs that showed anti-inflammatory effect in these studies is metformin (Han et al., 2018).

Metformin is an oral anti-diabetic drug from the class of biguanides. It is the first line treatment of diabetes type 2. It is widely used as it has good safety profile, low side effect and cheap cost (Malik et al., 2018). Studies have shown that metformin modulates cellular metabolism by two inter-related mechanisms. It transiently inhibits mitochondrial complex I of the electron transport chain, decreasing the production of mitochondrial reactive oxygen species and complex I inhibition also leads to an increase of the adenosine monophosphate/adenosine triphosphate (ATP) ratio (a critical signal of energy imbalance), which activates the AMPK. AMPK is a ubiquitous, critical cellular energy sensor with pleiotropic effects on cell metabolism, which can protect the cell by shutting down ATP consuming processes, promoting fatty acid oxidation and controlling the turn-over cycle of injured mitochondria. Metformin and AMPK activation improve endothelial function, reducing capillary leak and inducible nitric oxide synthase and increasing endothelial nitric oxide synthase activity potentially improving vascular tone and microvascular function (Gómez et al., 2022) Metformin has been reported to have an anti-inflammatory effect. In a prospective study to investigate the anti-inflammatory effect of AMPK activation in vivo, metformin and AICAR was administered respectively to mice prior to LPS injection. LPS injection significantly increased the level of VCAM1 in the arterioles, peritubular capillaries, post capillary venules, and glomerulus in the kidneys as well as in the arterioles, alveolar capillaries, and venules in the lungs. Metformin and AICAR administration effectively reduced VCAM1 expression in the microvascular beds both in the kidneys and lungs. Furthermore, LPS-induced increase of the serum levels of pro-inflammatory cytokines TNF⍺ and IL-6 were both significantly decreased by metformin and AICAR (Tian et al., 2019). In a trial of patients receiving glucocorticoid treatment for various chronic inflammatory diseases, 12 weeks of treatment with metformin 2550 mg/day resulted in lower serum levels of high-sensitive CRP as compared to placebo. Furthermore, carbohydrate-challenged TNF-α levels increased significantly in the placebo-treated group but not in the metformin-treated group (Pernicova et al., 2020) In addition, metformin showed some antibacterial activity. A retrospective study conducted in 2022 has shown that at the cellular level, metformin modulates cell metabolism through transient inhibition of complex I of mitochondrial electron transport chain and activates AMPK that protects energy balance in the cell (Gómez et al., 2022). It enhances neutrophil chemotaxis and phagocytosis and bacterial clearance (Bai and Chen, 2021).

Some studies have shown that metformin has a beneficial effect in sepsis patients. In two retrospective studies of septic shock patients receiving metformin, it showed an improvement in inflammatory response and oxidative stress induced by sepsis which resulted in improved mortality at different doses of metformin (Gras et al., 2006; Doenyas-Barak et al., 2015) . In a systematic review and meta-analysis done by Liang et al for published observational cohort data to determine the association between preadmission metformin use and mortality in septic adult patients with diabetes mellitus, it was concluded that preadmission metformin users had lower mortality than non-users and this analysis suggested that the effect of metformin is related to its anti-inflammatory effect (Liang et al., 2019).

Metformin has not significant adverse effects; however, it may cause gastrointestinal upset that can be overcome by titration of the dose and administration with meals (Nasri and Rafieian-Kopaei, 2014) and a rare but serious condition called lactic acidosis with the following symptoms: dizziness, severe drowsiness, muscle pain, tiredness, chills, blue/cold skin, fast/difficult breathing, slow/irregular heartbeat, stomach pain with diarrhea, nausea or vomiting. Lactic acidosis usually occurs due to drug overdose or in some contraindicated conditions (Scheen and Paquot, 2013). Rare incidence of lactic acidosis has been reported with the use of metformin especially in patients with renal impairment, hence, metformin is contraindicated in those with creatinine clearance less than 45ml/min. In sepsis, previous study reported that patients hospitalized for suspected sepsis who were on metformin had slightly higher prevalence of hyperlactatemia than non- metformin users though non-metformin users were found to have a higher 28-days mortality risk than metformin users (Green et al., 2012). In another study, conducted to compare the prognosis of extremely elevated plasma lactate levels and septic shock between metformin users and non-users it was found that the rate of in hospital mortality was lower for those who were actively treated with metformin than those who were not. the prognosis of metformin users were better despite higher lactate levels (Doenyas-Barak et al., 2015). One last study was done to evaluate the impact of metformin use on lactate kinetics in septic patients and showed that lactate levels in metformin users were initially elevated in the early phase in severe sepsis and septic shock. However, there was no significant difference in lactate levels, lactate clearance and normalization over the initial 24 hours period based on metformin use (Park et al., 2017)

To the best of our knowledge our study will be the first prospective controlled randomized trial to assess the clinical outcome of metformin in patients with sepsis.

ELIGIBILITY:
Inclusion Criteria:

* Age more than 18 years old.
* A diagnosis of sepsis according to the latest Sepsis-3 definition
* Estimated GFR >45 ml/min

Exclusion Criteria:

* • Immunosuppressed or end stage cancer.

  * Septic Shock.
  * Pregnancy and breast feeding.
  * Patients on metformin, Sodium glucose cotransporters or Gliptins.
  * End stage hepatic disease.
  * Contraindications to metformin (chronic respiratory failure, chronic cardiac failure, chronic kidney or liver disease, myocardial infarction within the last month).
  * Patients with hypersensitivity to metformin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2023-09-10 (Actual); Primary Completion 2024-06-15 (Estimated); Study Completion 2024-07-10 (Estimated)

PRIMARY OUTCOMES:
28 days mortality | 28 days
  Patients mortality rate and time from ICU admission till death due to any cause will be assessed within 28 days even after discharge from the ICU.

SECONDARY OUTCOMES:
2.Total ICU lengths of stay: | 28 days
  The number of days that the patient will stay in the ICU will be calculated.
3.Arterial blood gases (ABG): | 28 days
  ABG will be measured daily for every patient throughout his/her stay in the ICU. The total number of days that ABG are abnormal will be calculated for every patients in order to get the number of abnormal readings and check after how long ABG returned to normal
4- Serum TNF alpha: | 28 days
  Blood samples will be withdrawn at baseline and day ten of ICU admission from every patient included in the study to measure TNF alpha. Samples will be stored in -80C and will be assessed using ELISA technique.
5- Total Leucocytic Count (TLC): | 28 days
  Blood samples will be withdrawn daily from every patient included in the study to measure TLC. The total number of days that TLC is high will be calculated for every patients in order to get the number of abnormal readings and check after how long TLC returned to normal ( 4000 to 11,000/microliters).
6- Sequential organ Failure assessment Scores (SOFA): | 28 days
  SOFA score will be calculated daily for every patient to assess organ failure and recovery. Sequential Organ Failure Assessment score (SOFA) is a scoring system used to evaluate organ failure. The score is based on six different scores: respiratory, cardiovascular, hepatic, coagulation, renal and neurological system. It calculates the degree of organ failure by assigning a point of 0 (normal) to 4 (failure) for each organ. Score ranges from 0 (best) to 24 (worst) points. For calculating SOFA score the below table 1 will be used:(Singer et al., 2016a)
7- APACHE II Score: | 28 days
  APACH II score will be calculated daily for every patient to assess disease severity. The score can help in the assessment of patients to determine the level & degree of diagnostic & therapeutic intervention. Score ranges from minimum 0 and maximum 71; increasing score is associated with an increasing risk of hospital death. For calculating APACHE score, below table will be used (Akavipat, 2019)
8-GCS Score: | 28 days
  Glasgow Coma scale (GCS) will be calculated daily to assess patient's consciousness. It is scored between 3 and 15, with 3 being the worst and 15 the best. It is composed of 3 parameters: best eye response (E), best verbal response (V), and best motor response (M). A score of 13 or higher correlates with mild brain injury, a score of 9 to 12 correlates with moderate injury, and a score of 8 or less represents severe brain injury (Teasdale and Jennett, 1974).
9-28 days Readmission: | 28 days
  The number of patients who were discharged from the ICU and returned again within 28 days will be calculated
10-Blood Pressure | 28 days
  All patients included in the study will be monitored 24 hours a day (24/24) by putting them on a vital signs monitor in order to follow up their blood pressure. The total number of abnormal blood pressure measurements will be calculated for every patient. Mean arterial blood pressure will also be calculated (target is 65 mm Hg) and the total number of days patient will need a vasopressor will be calculated and doses of vasopressor will be documented.
11-Mechanical Ventilation: | 28 days
  Number of patients who will need mechanical ventilation will be calculated. In addition, ventilation free days will be assessed for every patient.
12-Serum Lactate levels: | 28 days
  Blood samples will be withdrawn every other day from every patient included in the study to measure serum lactate levels. The lactate cutoffs determining an elevated level ranged from 1.6-2.5 mmol/L (Evans et al., 2021). Patients with elevated serum lactate levels will be closely monitored. The number of days that serum lactate levels are high will be calculated for every patient throughout the study
GIT Disturbances: | 28 days
  Patient will be interviewed for the incidence of nausea, vomiting or diarrhea. If patient cannot reply (low conscious level), nurses will be asked. The total number of days that patient will suffer any of the GIT disturbances will be calculated and documented.

CONTACTS AND LOCATIONS:
Locations (1):
- Al Demerdash University Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No